CLINICAL TRIAL: NCT03443817
Title: Feasibility and Effect of a Follow up Tele-rehabilitation Program for Chronic Obstructive Lung Disease vs. Standard Follow up
Acronym: 2-TELEKOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Eurostars (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2-KOL
Record Dates: First submitted 2018-02-19; First posted 2018-02-23 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Feasibility; tele-rehabilitation; follow-up; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled trial comparing the effects of a follow-up tele-rehabilitation program and conventional follow-up rehabilitation in patients with severe COPD. 54 patients fulfilling the inclusion criteria will be randomized in two groups to either an 8 week follow-up tele-rehabilitation program or to standard follow up after rehabilitation. Participants will be tested at baseline, after 8 weeks and 6 months after cessation of the training programs. In the intervention group, a real- and a virtual physiotherapist agent will facilitate the rehabilitation.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): There is no conventional rehabilitation follow up program, but all patients are encouraged to continue training
- Intervention group (Experimental): The intervention group will obtain telerehabilitation
  Interventions: Behavioral: Tele rehab

INTERVENTIONS:
Behavioral: Tele rehab — Video Consultation (VC) Sessions: Each patient will have the opportunity to have minimum one VC per week the first month, one VC each second week the second month one VC a month
  Retraining breath: Patients will also be instructed to use different techniques to breath during the video consultations with the physiotherapist.
  Chat Sessions: Each patient has the opportunity to chat with the physiotherapist any time via the chat module of the system.
  Workout Sessions with a Virtual Physiotherapist Agent (VPA): The patient will train according to what is decided by the physiotherapist and the patient in the VC or chat meetings. Normally, the patients will train 10-20 minutes daily at home with its individual and tailored VPA.
  Patients' security: In order to minimize the risks of possible accidents while performing the exercises, the patient will answer questions before and after each exercise performance that the physiotherapist can follow in real time.
  Arms: Intervention group

SUMMARY:
Introduction In order to guarantee chronic patients & elderly a high quality service from health care organizations in the coming decades, new technologies have been implemented to treat patients from a distance. There is still a need for more studies on the efficacy and cost-effectiveness of tele-rehabilitation (TR) and its long-term effects needs also to be determined. To guarantee individuals with chronic obstructive pulmonary diseases (COPD) a high quality service from health care organizations in the coming decades and economically save the national health systems for an expensive bill for the treatment of COPD, new actions plans has to be taken into use. Hereby, more patients can be treated with less human resources while still sustaining or even improving today's services. The importance of such welfare action plans has to maintain a high quality of service that individuals with COPD are willing to accept. Here, TR seems to be a good welfare action plans. Despite proof of improved cost-effectiveness, no studies support the benefits of TR in COPD patient with respect to adherence, security, treatment efficacy and improved quality of life.

Aim To assess and compare the feasibility and effect of a tele-rehabilitation program with a new and innovative TR platform (NITRP) compared to standard treatment with respect to exercise capacity, quality of life and activities of daily living in patients with COPD.

Method and material The study is a prospective randomized controlled trial comparing the effects of a follow-up tele-rehabilitation program and conventional follow-up rehabilitation in patients with severe COPD. 54 patients fulfilling the inclusion criteria will be randomized in two groups to either an 8 week follow-up tele-rehabilitation program or to standard follow up after rehabilitation. Participants will be tested at baseline, after 8 weeks and 6 months after cessation of the training programs. In the intervention group, a real- and a virtual physiotherapist agent will facilitate the rehabilitation.

Ethical considerations This study will not pose any risk to the patient as compared to current practice. Participation is voluntary and the patient may at any time withdraw from the study without consequences for future care or treatment. The questionnaires and the test methods used are clinically recognized instruments. Signed informed consent will be obtained from the all participants after verbal and written information and before the study starts. The study will not be initiated before approval from the Ethics Committee and the Data Protection Agency has been obtained. The study will follow the general research ethical rules as expressed in the Helsinki Declaration II.

DETAILED DESCRIPTION:
Intro

To guarantee chronic patients and elderly a high quality service from health care organizations in the coming decades, new technologies has been implemented to treat patients from a distance. This document reflects the latest research studies based on tele-rehabilitation (TR), its application in chronic lung diseases and the topics that still needs to be investigated.

TR Studies of TR in patients with lymphedema (Galiano-Castillo et al., 2014) or COPD (Paneroni et al., 2014)(Tousignant et al., 2012)(Dinesen, Seeman, and Gustafsson, 2011)(Dinesen, Huniche, and Toft, 2013) or in the orthopedic areas as, lower back (Palacín-Marín et al., 2013), knee (Cabana et al., 2010) (Tousignant, Moffet, et al., 2011) (Tousignant, Boissy, et al., 2011) and shoulder (Eriksson et al., 2009)(Eriksson, Lindström and Ekenberg, 2011) show that tele-technology has been developed to a level where it is possible to treat, test and follow-up patients from a distance. Patients who have not been offered such solutions face increased risks of hospital-acquired infections (Dancer, 2009) and longer travel and waiting time to get treated. The public sector expects higher expenditure due to treatment and transportation cost, specifically in chronic patients and the elderly whose numbers tends to increase according to demographics trend (Palacín-Marín et al., 2013)(Barros et al., 2011)(Parker and Thorslund, 2007)(Yach, Hawkes, Gould, and Hofman, 2004). Such facts points to the need of creating and improving solution that overcome such health care challenges.

TR seems to be a good approach to reach patients in low inhabited areas (Hill and Sppath, 2010), changing health care to self-care (Haarder, 2011), empowering patient's awareness on their disease and increasing the flexibility patients need to acquire to obtain healthier behaviors. Although the interest in TR research is high, there is still a need for more studies on the efficacy (Paneroni et al., 2014) and cost-effectiveness of TR (Paneroni et al., 2014) (Langberg, Lindahl, Kidholm, and Dinesen, 2014) just as the long-term effects of TR have to be determined (Langberg et al., 2014).

Chronic obstructive pulmonary disease (COPD) COPD is among the most resource costly diseases we face in our century (Kjøller, Juel and Kamper-Jørgensen, 2007). In Denmark, approximately 430,000 people have COPD of which around 50,000 have severe COPD (Kirkegaard N, Brandt A, Timm H, 2013)(Mannino, Doherty and Sonia Buist, 2006). Eriksen (Eriksen and Vestbo, 2010) states that up to 42.3% of patients with COPD discharged from hospitals are readmitted the following year, and 17% of patients treated in emergency departments require hospitalization. Danish pulmonary physicians concluded that COPD cost the Danish society three billion DKK in 2002 (Hos, 2007) where up to 20% of the most severe COPD patients consume over 70% of the total health expenditure (Jansson et al., 2002). Nowadays, some municipalities have already problems with offering rehabilitation services to all COPD patients in some areas in Denmark (Kjøller, Juel and Kamper-Jørgensen, 2007). Actions implementing TR for COPD patients have been started and research begins to show some improvements.

Pulmonary rehabilitation in COPD The objective of treatment for patients with COPD is to delay the progression of the disease, prevent acute exacerbations, improve quality of life, reduce symptoms and reduce mortality. Rehabilitation of COPD includes among others physical training and patient education (Sundhedsstyrelsen, 2007). There is a need for an improved prevention and treatment of exacerbations (Barnes et al., 2013). Despite the poor evidence about determinants of physical activity and impact of treatment in COPD patients (Gimeno-Santos et al., 2014), a wide range of interventions are commonly used by physiotherapist to treat individuals with COPD (Kozu et al., 2011),(Kenn, Gloeckl and Behr, 2013) (Garrod and Lasserson, 2007). Researchers have shown significant improvement in general condition (Lacasse, Guyatt and Goldstein, 1997)(Ries et al., 1995)(Lacasse et al., 2009)(Nava, 1998)(Simpson et al., 1992), quality of life (Wijkstra et al., 1995)(Bendstrup et al., 1997), long-term survival (Godoy, 2007), sputum clearance (Garrod and Lasserson, 2007) (Oldenburg et al., 1979); Health-related quality of life (Almagro and Castro, 2013) (Blackstock et al., 2013) (Jones, 2013)(Bendstrup et al., 1997), training of muscle strength and exercise tolerance (Ortega et al., 2002)(Bendstrup et al., 1997), walking distance (Ries et al., 2007) (Ringbaek et al., 2008) (Wedzicha et al., 1998), exercise capacity, endurance (Lacasse, Guyatt and Goldstein, 1997) (Ries et al., 1995) (Lacasse et al., 2009) (Nava, 1998) (Simpson et al., 1992); days of hospitalization (Ries et al., 2007) (Griffiths et al., 2000), tachypnea (Lacasse, Guyatt and Goldstein, 1997) (Ortega et al., 2002) and morbidity (Godoy, 2007). Although the advantages of PR are many, its implementation should be placed alongside the routine treatment options (Ozalevli et al., 2010). It has been shown that the frequency of emergency department presentations and hospital admissions in COPD patients was significantly reduced after participation in early discharge care with ongoing follow-up support (Lawlor et al., 2009).

Tele-rehabilitation in COPD Tele-rehabilitation at home is feasible and well accepted by patients, although technology may be perceived as difficult (Paneroni et al., 2014)(Tousignant et al., 2012). It seems to improve walking capacity, dyspnea, quality of life and daily physical activity (Paneroni et al., 2014). The interaction between the COPD patients at home and the healthcare professionals at the clinic through TR has evolved as a dialogue channel forming the basis for mutual learning processes and new relationships (Dinesen et al., 2011). Here, patients exhibit four types of attitudes about their tele-rehabilitation: indifference, learning as part of situations in everyday life, feeling of security and motivation for performing physical training (Dinesen, Huniche and Toft, 2013). Preliminary evaluations from tele-rehabilitation initiatives in Scotland showed tele-rehabilitation to be more cost effective for patients living in remote areas compared to an out-reach- or centralized model (Hill and Sppath, 2010).

Hypothesis:

There is still a need for more studies of the efficacy and cost-effectiveness of TR, just as also the long-term effects of TR have to be determined. To guarantee individuals with COPD a qualitative service from health care organizations in the coming decades and economically save the national health systems for an expensive bill to treating COPD, new actions plans has to be taken in mind in order to treat more patients with less human resources and still sustaining or improving today's services. The importance of such welfare action plans has to maintain a quality of service that individuals with COPD are willing to accept. Here, TR seems to be a good welfare action plans. Despite improved cost effectiveness, evidence supporting patient ´s adherence and security, treatment efficacy and improvements of quality of life with tele-rehabilitation in COPD is still warranted.

To assess and compare the feasibility and effect of a follow-up tele-rehabilitation program after standard COPD rehabilitation with a new and innovative TR platform (NITRP) compared to standard follow-up after COPD rehabilitation with respect to exercise capacity, quality of life and activities of daily living in patients with COPD.

The primary purpose of the study is to assess the effect of tele-rehabilitation after standard COPD rehabilitation with a NITRP compared to the usual follow-up after standard COPD rehabilitation on exercise capacity and quality of life in COPD patients based on the following hypotheses:

Activities of daily living, exercise capacity and health-related quality of life are equal or improved by follow-up tele-rehabilitation after standard COPD rehabilitation compared to follow-up.

The secondary purpose is to investigate the efficacy and cost effectiveness of follow-up tele-rehabilitation after standard COPD rehabilitation with a NITRP compared to usual follow-up on "number of acute exacerbations and number of visits to the health care system in a period of time" and "rehabilitation- and transportation costs" in rehabilitation of COPD patients based on the following hypothesis:

The rehabilitation costs of tele-rehabilitation after standard COPD rehabilitation are lower or equal compared to conventional rehabilitation response.

ELIGIBILITY:
Inclusion Criteria:

1. Stable COPD
2. Signed informed consent
3. Completion of the standard rehabilitation program
4. Permanent oxygen therapy is not an obstacle for participation.

Exclusion Criteria:

1. The patient has significant musculoskeletal disorders that limit his / her function levels to a degree that is not caused by dyspnea
2. The patient has pronounced dizziness, significant sensory or motor disability, dementia or terminal malignant disease
3. Serious comorbidities (unstable heart disease, irregular diabetes, known malignant disease, another disease that makes the patient unfit to participate in the study).
4. Non-compliant patient (eg. Nursing Homes Residents)
5. Participation in another project within the last 30 days
6. Mini-Mental State Examination score less than 24 points
7. Severe vision or hearing loss.
8. Non-Danish speaking.
9. Lack of will to implement the protocol.
10. Motor or sensory disease, which makes it impossible for walk training
11. Have experienced a worsening in the last 4-6 weeks
12. Musculoskeletal disorders
13. Serious heart diseases (ejection fraction <30%, daily angina, or as indicated by treating the cardiologist)
14. Can not understand informed consent
15. Other factors that inhibit the use of telerehabilitation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test | measured at week 8
  Change in the 6 minute walk test

SECONDARY OUTCOMES:
6 minute walk test | 6 months after cessation
  Change in the 6 minute walk test measured 6 months after cessation of the tele-rehabilitation program compared to baseline.
Health-related quality of life | 8 weeks, and 6 months after cessation
  Change in total score in health-related quality of life measured by SGRQ after 8 weeks, and 6 months after cessation of the tele-rehabilitation program compared to baseline.
Generalised Anxiety Disorder Assessment (GAD-7) | 8 weeks, and 6 months after cessation
  Change in total score in health-related quality of life measured by GAD-7 after 8 weeks, and 6 months after cessation of the tele-rehabilitation program compared to baseline.
  The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
health-related quality of life measured by SGRQ | 6 months after cessation
  Change in component scores (symptoms, activity & impact) in health-related quality of life measured by SGRQ immediately after, and 6 months after cessation of the tele-rehabilitation program compared to baseline.
Cost tele-rehab | 6 months
  Cost of the tele-rehabilitation program

CONTACTS AND LOCATIONS:
Overall Officials: Jose Cerdan, Principal Investigator — Aarhus University Hospital
Locations (1):
- Jose Cerdan, Aarhus, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
The study is approved by the Data Protection Agency for permission for data recording and storage of data. The data will be rendered anonymous through a code system and stored safely in accordance with applicable rules of the organizers. The study follows the general research ethics rules as expressed in the Helsinki Declaration II ('World Medical Association Declaration of Helsinki: Ethical Principles for Medical Research involving Human Subjects', 2000).

REFERENCES:
- [Background] Tsai LL, McNamara RJ, Moddel C, Alison JA, McKenzie DK, McKeough ZJ. Home-based telerehabilitation via real-time videoconferencing improves endurance exercise capacity in patients with COPD: The randomized controlled TeleR Study. Respirology. 2017 May;22(4):699-707. doi: 10.1111/resp.12966. Epub 2016 Dec 19. PMID 27992099
- [Background] Zanaboni P, Dinesen B, Hjalmarsen A, Hoaas H, Holland AE, Oliveira CC, Wootton R. Long-term integrated telerehabilitation of COPD Patients: a multicentre randomised controlled trial (iTrain). BMC Pulm Med. 2016 Aug 22;16(1):126. doi: 10.1186/s12890-016-0288-z. PMID 27549782
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633